CLINICAL TRIAL: NCT02611362
Title: A Multilevel Gaming Intervention for Persons on PrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Laura Whiteley, Co-Director, Young Adult Behavioral Health, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R34MH104068 (NIH)
Record Dates: First submitted 2015-11-03; First posted 2015-11-20 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: MSM; PrEP; HIV Risk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Subjects in the intervention group will each receive a smartphone with a data service plan as the active arm. The IMB Gaming Intervention is designed to improve information, motivation, and skills about adherence and HIV preventative behaviors throughout play. The mission of Viral Combat is: kill virus and build strength through taking medicine, learning HIV prevention information, and engaging with healthy characters in order to improve motivation and build skills. Participants will get a game graphic with a supportive message such as "Missing you: Get in the Game" to their phones. Throughout the gaming intervention subjects will continue routine clinical care visits and HIV testing in the PrEP clinic.
  Interventions: Behavioral: IMB Gaming Intervention
- Comparison (No Intervention): This condition will be matched with the IMB Gaming Intervention for appeal, time and attention. Subjects in COMP will each receive smartphones with the same data service plan as the active arm. Smartphones given to participants in COMP will have a stylistically similar non-PrEP, non-IMB game designed by Mission Critical Studios (Dr. Nano X: Incredible Voyage Inside The Body, http://www.youtube.com/watch?v=lyHzSZFzU1Q ). This is the same game that Viral Combat is being adapted from. Therefore, the iPhone game in COMP will have a look and feel that is very similar to our intervention game but without IMB, PrEP, and HIV prevention related content. Similar to the Intervention group, participants will have routine clinical care visits in the PrEP clinic (or more frequently if needed for urgent care).

INTERVENTIONS:
Behavioral: IMB Gaming Intervention
  Arms: Intervention

SUMMARY:
This study will develop and test a novel, smartphone based gaming intervention to improve adherence to medication to prevent HIV (known as Pre-exposure Prophylaxis, PrEP) and to decrease HIV risk behaviors among men who have sex with men (MSM). In the intervention, participants will engage with an immersive app/game on their iPhone. While gaming, participants will gain information about their health, improve motivation for PrEP and medical appointment adherence, and practice healthy behaviors. If the intervention is found to be effective, it can be tested in a larger study and then disseminated to other people taking PrEP.

DETAILED DESCRIPTION:
The use of antiretroviral medications to reduce the risk of acquiring HIV infection (Pre-exposure Prophylaxis, PrEP) is an efficacious and promising new prevention strategy. In published studies, failure of PrEP was associated with poor adherence and low plasma drug levels. This indicates that optimal PrEP treatment will require behavioral interventions to promote adherence. Averting increases in risk behavior will also be essential for maintaining PrEP's protective effects. Interventions will need to address on-going HIV risk behavior and be relevant for persons using PrEP (e.g. young adult MSM). Borrowing from recent literature in HIV prevention and treatment adherence, interventions that utilize intuitive easy to use technologies with motivational components show promise for behavior change and dissemination.

This study will examine an interactive smartphone based app/game that is immersive and appealing. This novel, but intuitive multi-level technology will measure PrEP adherence, promote engagement in treatment and safe sexual behavior. The smartphone app/game will be developed to include content consistent with the Information-Motivation-Behavioral Skills (IMB) Model. While gaming, participants will experience absorbing action-oriented adventures that increase information about their health (e.g. knowledge about PrEP treatment and HIV), improve motivation (e.g. action-figures experience health benefits of adherence), and build skills (e.g. utilize clinicians as partners, condom self efficacy). In-depth interviews with young adults on PrEP and an open trial of the intervention will inform the development of the intervention and procedures. A small randomized controlled pilot study among 50 participants on PrEP will examine the preliminary efficacy of the intervention (IMB informed app/game). It is hypothesized that, compared to subjects in the control group, participants in the IMB Gaming Intervention will show: improved adherence to PrEP, higher blood ARV levels, decreased HIV risk behaviors, and improved self efficacy and attitudes for PrEP treatment adherence.

The specific aims are:

1. To create an engaging and absorbing smartphone based app/game with content consistent with the Information-Motivation-Behavioral Skills (IMB) model to measure and improve PrEP treatment adherence and safer sex behaviors, and to receive feedback on the game's utility and acceptability from in-depth interviews with MSM (estimated mean age 27).
2. To conduct an open trial of the IMB Gaming Intervention with MSM to obtain further qualitative and quantitative information on its acceptability, and feasibility. These data will be used to modify the approach and technology as needed.
3. To evaluate, in a 24 week randomized controlled pilot study (n=50), the preliminary efficacy of the IMB Gaming Intervention compared to a time, attention, and technology matched group. Investigators will examine the impact of the IMB Gaming Intervention in improving treatment adherence (measured by clinic visits attended, self-report) and biological measures (ARV levels). Investigators will also examine the impact on HIV risk behaviors.

ELIGIBILITY:
Inclusion Criteria: All males on PrEP over the age of 18

* English speaking
* Receiving prophylactic antiretroviral treatment
* Not enrolled in another PrEP related study
* Able to give consent/assent and not impaired by cognitive or medical limitations as per clinical assessment.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Whiteley, MD, Principal Investigator — Brown University
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Background] Underhill K, Operario D, Skeer M, Mimiaga M, Mayer K. Packaging PrEP to Prevent HIV: An Integrated Framework to Plan for Pre-Exposure Prophylaxis Implementation in Clinical Practice. J Acquir Immune Defic Syndr. 2010 Sep;55(1):8-13. doi: 10.1097/qai.0b013e3181e8efe4. PMID 21423876
- [Background] Padian NS, Buve A, Balkus J, Serwadda D, Cates W Jr. Biomedical interventions to prevent HIV infection: evidence, challenges, and way forward. Lancet. 2008 Aug 16;372(9638):585-99. doi: 10.1016/S0140-6736(08)60885-5. Epub 2008 Aug 5. PMID 18687456
- [Background] UNAIDS. Global Facts & Figures. Geneva, Switzerland: Joint United Nations Programme on HIV/ AIDS; 2012.
- [Background] Szekeres G, Coates TJ. Policy and practice implications of HIV pre-exposure prophylaxis (PrEP) in the United States. Los Angeles, CA: UCLA Program in Global Health, AIDS Policy Development Center; 2006.
- [Background] Paxton LA, Hope T, Jaffe HW. Pre-exposure prophylaxis for HIV infection: what if it works? Lancet. 2007 Jul 7;370(9581):89-93. doi: 10.1016/S0140-6736(07)61053-8. No abstract available. PMID 17617276
- [Background] Abdool Karim SS. Antiretroviral chemoprophylaxis for the prevention of HIV infection: future implementation challenges. HIV Therapy. 2009; 3(1):3-6.
- [Background] CDC. Pre-exposure prophylaxis (PrEP) for HIV prevention: planning for potential implementation in the U.S. Atlanta, GA: 2009
- [Background] Rotheram-Borus MJ, Swendeman D, Chovnick G. The past, present, and future of HIV prevention: integrating behavioral, biomedical, and structural intervention strategies for the next generation of HIV prevention. Annu Rev Clin Psychol. 2009;5:143-67. doi: 10.1146/annurev.clinpsy.032408.153530. PMID 19327028
- [Background] Liu AY, Grant RM, Buchbinder SP. Preexposure prophylaxis for HIV: unproven promise and potential pitfalls. JAMA. 2006 Aug 16;296(7):863-5. doi: 10.1001/jama.296.7.863. No abstract available. PMID 16905792
- [Background] Mayer KH, Wheeler DP, Bekker LG, Grinsztejn B, Remien RH, Sandfort TG, Beyrer C. Overcoming biological, behavioral, and structural vulnerabilities: new directions in research to decrease HIV transmission in men who have sex with men. J Acquir Immune Defic Syndr. 2013 Jul;63 Suppl 2(0 2):S161-7. doi: 10.1097/QAI.0b013e318298700e. PMID 23764630
- [Background] Paltiel AD, Freedberg KA, Scott CA, Schackman BR, Losina E, Wang B, Seage GR 3rd, Sloan CE, Sax PE, Walensky RP. HIV preexposure prophylaxis in the United States: impact on lifetime infection risk, clinical outcomes, and cost-effectiveness. Clin Infect Dis. 2009 Mar 15;48(6):806-15. doi: 10.1086/597095. PMID 19193111
- [Background] Abbas UL, Anderson RM, Mellors JW. Potential impact of antiretroviral chemoprophylaxis on HIV-1 transmission in resource-limited settings. PLoS One. 2007 Sep 19;2(9):e875. doi: 10.1371/journal.pone.0000875. PMID 17878928
- [Background] Desai K, Sansom SL, Ackers ML, Stewart SR, Hall HI, Hu DJ, Sanders R, Scotton CR, Soorapanth S, Boily MC, Garnett GP, McElroy PD. Modeling the impact of HIV chemoprophylaxis strategies among men who have sex with men in the United States: HIV infections prevented and cost-effectiveness. AIDS. 2008 Sep 12;22(14):1829-39. doi: 10.1097/QAD.0b013e32830e00f5. PMID 18753932
- [Background] Golub SA, Kowalczyk W, Weinberger CL, Parsons JT. Preexposure prophylaxis and predicted condom use among high-risk men who have sex with men. J Acquir Immune Defic Syndr. 2010 Aug;54(5):548-55. doi: 10.1097/QAI.0b013e3181e19a54. PMID 20512046
- [Background] Amico KR, Mansoor LE, Corneli A, Torjesen K, van der Straten A. Adherence support approaches in biomedical HIV prevention trials: experiences, insights and future directions from four multisite prevention trials. AIDS Behav. 2013 Jul;17(6):2143-55. doi: 10.1007/s10461-013-0429-9. PMID 23435697
- [Background] Baeten JM, Donnell D, Ndase P, Mugo NR, Campbell JD, Wangisi J, Tappero JW, Bukusi EA, Cohen CR, Katabira E, Ronald A, Tumwesigye E, Were E, Fife KH, Kiarie J, Farquhar C, John-Stewart G, Kakia A, Odoyo J, Mucunguzi A, Nakku-Joloba E, Twesigye R, Ngure K, Apaka C, Tamooh H, Gabona F, Mujugira A, Panteleeff D, Thomas KK, Kidoguchi L, Krows M, Revall J, Morrison S, Haugen H, Emmanuel-Ogier M, Ondrejcek L, Coombs RW, Frenkel L, Hendrix C, Bumpus NN, Bangsberg D, Haberer JE, Stevens WS, Lingappa JR, Celum C; Partners PrEP Study Team. Antiretroviral prophylaxis for HIV prevention in heterosexual men and women. N Engl J Med. 2012 Aug 2;367(5):399-410. doi: 10.1056/NEJMoa1108524. Epub 2012 Jul 11. PMID 22784037
- [Background] Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV; iPrEx Study Team. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med. 2010 Dec 30;363(27):2587-99. doi: 10.1056/NEJMoa1011205. Epub 2010 Nov 23. PMID 21091279
- [Background] Thigpen MC, Kebaabetswe PM, Paxton LA, Smith DK, Rose CE, Segolodi TM, Henderson FL, Pathak SR, Soud FA, Chillag KL, Mutanhaurwa R, Chirwa LI, Kasonde M, Abebe D, Buliva E, Gvetadze RJ, Johnson S, Sukalac T, Thomas VT, Hart C, Johnson JA, Malotte CK, Hendrix CW, Brooks JT; TDF2 Study Group. Antiretroviral preexposure prophylaxis for heterosexual HIV transmission in Botswana. N Engl J Med. 2012 Aug 2;367(5):423-34. doi: 10.1056/NEJMoa1110711. Epub 2012 Jul 11. PMID 22784038
- [Background] Van Damme L, Corneli A, Ahmed K, Agot K, Lombaard J, Kapiga S, Malahleha M, Owino F, Manongi R, Onyango J, Temu L, Monedi MC, Mak'Oketch P, Makanda M, Reblin I, Makatu SE, Saylor L, Kiernan H, Kirkendale S, Wong C, Grant R, Kashuba A, Nanda K, Mandala J, Fransen K, Deese J, Crucitti T, Mastro TD, Taylor D; FEM-PrEP Study Group. Preexposure prophylaxis for HIV infection among African women. N Engl J Med. 2012 Aug 2;367(5):411-22. doi: 10.1056/NEJMoa1202614. Epub 2012 Jul 11. PMID 22784040
- [Background] Microbicide Trials Network. MTN statement on decision to discontinue use of oral Tenofovir tablets in VOICE, a major HIV prevention study in women. 2011. Available at: http://www.mtnstopshiv.org/node/3619. Accessed Sept 25 2011. (VOICES)
- [Background] Centers for Disease Control and Prevention (CDC). Interim guidance: preexposure prophylaxis for the prevention of HIV infection in men who have sex with men. MMWR Morb Mortal Wkly Rep. 2011 Jan 28;60(3):65-8. PMID 21270743
- [Background] Cassell MM, Halperin DT, Shelton JD, Stanton D. Risk compensation: the Achilles' heel of innovations in HIV prevention? BMJ. 2006 Mar 11;332(7541):605-7. doi: 10.1136/bmj.332.7541.605. PMID 16528088
- [Background] Kates J, Levi J. Insurance coverage and access to HIV testing and treatment: considerations for individuals at risk for infection and for those with undiagnosed infection. Clin Infect Dis. 2007 Dec 15;45 Suppl 4:S255-60. doi: 10.1086/522547. PMID 18190296
- [Background] World Health Organization. Priority interventions: HIV prevention, treatment, and care in the health sector. Geneva: World Health Organization HIV/AIDS Department; 2009.
- [Background] Hogben M, Liddon N. Disinhibition and risk compensation: scope, definitions, and perspective. Sex Transm Dis. 2008 Dec;35(12):1009-10. doi: 10.1097/OLQ.0b013e31818eb752. No abstract available. PMID 18936724
- [Background] Grant RM, Buchbinder S, Cates W Jr, Clarke E, Coates T, Cohen MS, Delaney M, Flores G, Goicochea P, Gonsalves G, Harrington M, Lama JR, MacQueen KM, Moore JP, Peterson L, Sanchez J, Thompson M, Wainberg MA. AIDS. Promote HIV chemoprophylaxis research, don't prevent it. Science. 2005 Sep 30;309(5744):2170-1. doi: 10.1126/science.1116204. No abstract available. PMID 16195446
- [Background] Schechter M, do Lago RF, Mendelsohn AB, Moreira RI, Moulton LH, Harrison LH; Praca Onze Study Team. Behavioral impact, acceptability, and HIV incidence among homosexual men with access to postexposure chemoprophylaxis for HIV. J Acquir Immune Defic Syndr. 2004 Apr 15;35(5):519-25. doi: 10.1097/00126334-200404150-00010. PMID 15021317
- [Background] Martin JN, Roland ME, Neilands TB, Krone MR, Bamberger JD, Kohn RP, Chesney MA, Franses K, Kahn JO, Coates TJ, Katz MH. Use of postexposure prophylaxis against HIV infection following sexual exposure does not lead to increases in high-risk behavior. AIDS. 2004 Mar 26;18(5):787-92. doi: 10.1097/00002030-200403260-00010. PMID 15075514
- [Background] Farr G, Acosta Castro LA, DiSantostefano R, Claassen E, Olguin F. Use of spermicide and impact of prophylactic condom use among sex workers in Santa Fe de Bogota, Colombia. Sex Transm Dis. 1996 May-Jun;23(3):206-12. doi: 10.1097/00007435-199605000-00008. PMID 8724510
- [Background] Roddy RE, Zekeng L, Ryan KA, Tamoufe U, Tweedy KG. Effect of nonoxynol-9 gel on urogenital gonorrhea and chlamydial infection: a randomized controlled trial. JAMA. 2002 Mar 6;287(9):1117-22. doi: 10.1001/jama.287.9.1117. PMID 11879108
- [Background] Crepaz N, Hart TA, Marks G. Highly active antiretroviral therapy and sexual risk behavior: a meta-analytic review. JAMA. 2004 Jul 14;292(2):224-36. doi: 10.1001/jama.292.2.224. PMID 15249572
- [Background] Shaw A. Putting the Gay in Games: Cultural Production and GLBT Content in Video Games. Games and Culture. 2009; 4(3):228-253.
- [Background] Lopez, V. Ms. Pac-Man's gay kids: The growing number of out video gamers has led to more gay game characters.The Advocate, 2004. [Accessed 5/11/07 from http://findarticles.com/ p/articles/mi_m1589/is_2004_Nov_23/ai_n8700526]
- [Background] Gay gamers push for more player choice, like same-sex smooching in'Bully'.MTV.com. [Accessed 7/13/13 from http://www.mtv.com/news/articles/1557022/20070412/index.jhtml
- [Background] Pew Internet and American Life. Two-thirds of young adults and those with higher income are smartphone owners. Washington, DC: Pew Internet & American Life Project; Sept 11, 2012. [Accessed 8/16/13 from http://pewinternet.org/~/media/Files/Reports/2012/PIP_Smartphones_Sept12%209%2010%2012.pdf]
- [Background] LGBT Market Research and Development Lab. The LGBT Community Survey. San Francisco, CA: Community Marketing Inc; 2012. [Accessed 5/12/12 from http://www.communitymarketinginc.com/documents/CMI_6th_LGBT_Community_Survey_USv1.pdf ]
- [Background] Horrigan J. Mobile access to data and information. Pew Internet and American Life Project. Pew Research Center. Mar 5, 2008. [Accessed 8/1/13 from: http://www.pewinternet.org/pdfs/PIP_Mobile.Data.Access.pdf]
- [Background] Mobile marvels: a special report on telecoms in emerging markets. The Economist. September 26, 2009. [Accessed 4/12/13 from http://www.economist.com/node/14483896]
- [Background] Swendeman D, Rotheram-Borus MJ. Innovation in sexually transmitted disease and HIV prevention: internet and mobile phone delivery vehicles for global diffusion. Curr Opin Psychiatry. 2010 Mar;23(2):139-44. doi: 10.1097/YCO.0b013e328336656a. PMID 20087189
- [Background] Esposito-Smythers C, Brown LK, Wolff J, Xu J, Thornton S, Tidey J; Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN 069). Substance abuse treatment for HIV infected young people: an open pilot trial. J Subst Abuse Treat. 2014 Feb;46(2):244-50. doi: 10.1016/j.jsat.2013.07.008. Epub 2013 Aug 27. PMID 23988190
- [Background] Carey MP, Schroder KE. Development and psychometric evaluation of the brief HIV Knowledge Questionnaire. AIDS Educ Prev. 2002 Apr;14(2):172-82. doi: 10.1521/aeap.14.2.172.23902. PMID 12000234
- [Background] Jaworski BC, Carey MP. Development and psychometric evaluation of a self-administered questionnaire to measure knowledge of sexually transmitted diseases. AIDS Behav. 2007 Jul;11(4):557-74. doi: 10.1007/s10461-006-9168-5. Epub 2006 Oct 3. PMID 17016760
- [Background] Eaton LA, Kalichman S. Risk compensation in HIV prevention: implications for vaccines, microbicides, and other biomedical HIV prevention technologies. Curr HIV/AIDS Rep. 2007 Dec;4(4):165-72. doi: 10.1007/s11904-007-0024-7. PMID 18366947
- [Background] Vanable PA, Carey MP, Brown JL, DiClemente RJ, Salazar LF, Brown LK, Romer D, Valois RF, Hennessy M, Stanton BF. Test-retest reliability of self-reported HIV/STD-related measures among African-American adolescents in four U.S. cities. J Adolesc Health. 2009 Mar;44(3):214-21. doi: 10.1016/j.jadohealth.2008.09.002. Epub 2008 Nov 20. PMID 19237106
- [Background] Saberi P, Johnson MO. Technology-based self-care methods of improving antiretroviral adherence: a systematic review. PLoS One. 2011;6(11):e27533. doi: 10.1371/journal.pone.0027533. Epub 2011 Nov 30. PMID 22140446
- [Background] Simoni JM, Frick PA, Pantalone DW, Turner BJ. Antiretroviral adherence interventions: a review of current literature and ongoing studies. Top HIV Med. 2003 Nov-Dec;11(6):185-98. PMID 14724327
- [Background] Haynes RB, Ackloo E, Sahota N, McDonald HP, Yao X. Interventions for enhancing medication adherence. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD000011. doi: 10.1002/14651858.CD000011.pub3. PMID 18425859
- [Background] Van Dyke RB, Lee S, Johnson GM, Wiznia A, Mohan K, Stanley K, Morse EV, Krogstad PA, Nachman S; Pediatric AIDS Clinical Trials Group Adherence Subcommittee Pediatric AIDS Clinical Trials Group 377 Study Team. Reported adherence as a determinant of response to highly active antiretroviral therapy in children who have human immunodeficiency virus infection. Pediatrics. 2002 Apr;109(4):e61. doi: 10.1542/peds.109.4.e61. PMID 11927734
- [Background] Watson DC, Farley JJ. Efficacy of and adherence to highly active antiretroviral therapy in children infected with human immunodeficiency virus type 1. Pediatr Infect Dis J. 1999 Aug;18(8):682-9. doi: 10.1097/00006454-199908000-00006. PMID 10462336
- [Background] Lima VD, Harrigan R, Murray M, Moore DM, Wood E, Hogg RS, Montaner JS. Differential impact of adherence on long-term treatment response among naive HIV-infected individuals. AIDS. 2008 Nov 12;22(17):2371-80. doi: 10.1097/QAD.0b013e328315cdd3. PMID 18981777
- [Background] Reisner SL, Mimiaga MJ, Skeer M, Perkovich B, Johnson CV, Safren SA. A review of HIV antiretroviral adherence and intervention studies among HIV-infected youth. Top HIV Med. 2009 Feb-Mar;17(1):14-25. PMID 19270345
- [Background] Bain-Brickley D, Butler LM, Kennedy GE, Rutherford GW. Interventions to improve adherence to antiretroviral therapy in children with HIV infection. Cochrane Database Syst Rev. 2011 Dec 7;2011(12):CD009513. doi: 10.1002/14651858.CD009513. PMID 22161452
- [Background] Samet JH, Horton NJ, Meli S, Dukes K, Tripps T, Sullivan L, Freedberg KA. A randomized controlled trial to enhance antiretroviral therapy adherence in patients with a history of alcohol problems. Antivir Ther. 2005;10(1):83-93. doi: 10.1177/135965350501000106. PMID 15751766
- [Background] Crankshaw T, Corless IB, Giddy J, Nicholas PK, Eichbaum Q, Butler LM. Exploring the patterns of use and the feasibility of using cellular phones for clinic appointment reminders and adherence messages in an antiretroviral treatment clinic, Durban, South Africa. AIDS Patient Care STDS. 2010 Nov;24(11):729-34. doi: 10.1089/apc.2010.0146. Epub 2010 Nov 1. PMID 21039181
- [Background] Safren SA, Hendriksen ES, Desousa N, Boswell SL, Mayer KH. Use of an on-line pager system to increase adherence to antiretroviral medications. AIDS Care. 2003 Dec;15(6):787-93. doi: 10.1080/09540120310001618630. PMID 14617500
- [Background] Simoni JM, Huh D, Frick PA, Pearson CR, Andrasik MP, Dunbar PJ, Hooton TM. Peer support and pager messaging to promote antiretroviral modifying therapy in Seattle: a randomized controlled trial. J Acquir Immune Defic Syndr. 2009 Dec 1;52(4):465-473. doi: 10.1097/qai.0b013e3181b9300c. PMID 19911481
- [Background] Andrade AS, McGruder HF, Wu AW, Celano SA, Skolasky RL Jr, Selnes OA, Huang IC, McArthur JC. A programmable prompting device improves adherence to highly active antiretroviral therapy in HIV-infected subjects with memory impairment. Clin Infect Dis. 2005 Sep 15;41(6):875-82. doi: 10.1086/432877. Epub 2005 Aug 5. PMID 16107989
- [Background] Wu AW, Snyder CF, Huang IC, Skolasky R, McGruder HF, Celano SA, Selnes OA, Andrade AS. A randomized trial of the impact of a programmable medication reminder device on quality of life in patients with AIDS. AIDS Patient Care STDS. 2006 Nov;20(11):773-81. doi: 10.1089/apc.2006.20.773. PMID 17134351
- [Background] Harris LT, Lehavot K, Huh D, Yard S, Andrasik MP, Dunbar PJ, Simoni JM. Two-way text messaging for health behavior change among human immunodeficiency virus-positive individuals. Telemed J E Health. 2010 Dec;16(10):1024-9. doi: 10.1089/tmj.2010.0050. Epub 2010 Nov 18. PMID 21087122
- [Background] Hugen PW, Langebeek N, Burger DM, Zomer B, van Leusen R, Schuurman R, Koopmans PP, Hekster YA. Assessment of adherence to HIV protease inhibitors: comparison and combination of various methods, including MEMS (electronic monitoring), patient and nurse report, and therapeutic drug monitoring. J Acquir Immune Defic Syndr. 2002 Jul 1;30(3):324-34. doi: 10.1097/00126334-200207010-00009. PMID 12131570
- [Background] Dunbar PJ, Madigan D, Grohskopf LA, Revere D, Woodward J, Minstrell J, Frick PA, Simoni JM, Hooton TM. A two-way messaging system to enhance antiretroviral adherence. J Am Med Inform Assoc. 2003 Jan-Feb;10(1):11-5. doi: 10.1197/jamia.m1047. PMID 12509353
- [Background] Paterson D, Swindells S, Mohr J, et al. How much adherence is enough? A prospective study of adherence to protease inhibitor therapy using MEMS caps. In: Program and abstracts of the 6th Conference on Retroviruses and Opportunistic Infections; January 31-February 4, 1999; Chicago. Abstract 92.
- [Background] Wise J, Operario D. Use of electronic reminder devices to improve adherence to antiretroviral therapy: a systematic review. AIDS Patient Care STDS. 2008 Jun;22(6):495-504. doi: 10.1089/apc.2007.0180. PMID 18462071
- [Background] Mannheimer SB, Morse E, Matts JP, Andrews L, Child C, Schmetter B, Friedland GH; Terry Beirn Community Programs for Clinical Research on AIDS. Sustained benefit from a long-term antiretroviral adherence intervention. Results of a large randomized clinical trial. J Acquir Immune Defic Syndr. 2006 Dec 1;43 Suppl 1:S41-7. doi: 10.1097/01.qai.0000245887.58886.ac. PMID 17091022
- [Background] Farmer KC. Methods for measuring and monitoring medication regimen adherence in clinical trials and clinical practice. Clin Ther. 1999 Jun;21(6):1074-90; discussion 1073. doi: 10.1016/S0149-2918(99)80026-5. PMID 10440628
- [Background] Arnsten JH, Demas PA, Farzadegan H, Grant RW, Gourevitch MN, Chang CJ, Buono D, Eckholdt H, Howard AA, Schoenbaum EE. Antiretroviral therapy adherence and viral suppression in HIV-infected drug users: comparison of self-report and electronic monitoring. Clin Infect Dis. 2001 Oct 15;33(8):1417-23. doi: 10.1086/323201. Epub 2001 Sep 5. PMID 11550118
- [Background] Smith SR, Brock TP, Howarth SM. Use of personal digital assistants to deliver education about adherence to antiretroviral medications. J Am Pharm Assoc (2003). 2005 Sep-Oct;45(5):625-8. doi: 10.1331/1544345055001292. No abstract available. PMID 16295649
- [Background] Kalichman SC, Rompa D, DiFonzo K, Simpson D, Austin J, Luke W, Kyomugisha F, Buckles J. HIV treatment adherence in women living with HIV/AIDS: research based on the Information-Motivation-Behavioral Skills model of health behavior. J Assoc Nurses AIDS Care. 2001 Jul-Aug;12(4):58-67. doi: 10.1016/S1055-3290(06)60217-3. PMID 11486721
- [Background] Levy RW, Rayner CR, Fairley CK, Kong DC, Mijch A, Costello K, McArthur C; Melbourne Adherence Group. Multidisciplinary HIV adherence intervention: a randomized study. AIDS Patient Care STDS. 2004 Dec;18(12):728-35. doi: 10.1089/apc.2004.18.728. PMID 15659884
- [Background] Golin CE, Liu H, Hays RD, Miller LG, Beck CK, Ickovics J, Kaplan AH, Wenger NS. A prospective study of predictors of adherence to combination antiretroviral medication. J Gen Intern Med. 2002 Oct;17(10):756-65. doi: 10.1046/j.1525-1497.2002.11214.x. PMID 12390551
- [Background] Fairley CK, Levy R, Rayner CR, Allardice K, Costello K, Thomas C, McArthur C, Kong D, Mijch A, Melbourne Adherence Group; Melbourne Adherence Group. Randomized trial of an adherence programme for clients with HIV. Int J STD AIDS. 2003 Dec;14(12):805-9. doi: 10.1258/095646203322556129. PMID 14678587
- [Background] Lyon ME, Trexler C, Akpan-Townsend C, Pao M, Selden K, Fletcher J, Addlestone IC, D'Angelo LJ. A family group approach to increasing adherence to therapy in HIV-infected youths: results of a pilot project. AIDS Patient Care STDS. 2003 Jun;17(6):299-308. doi: 10.1089/108729103322108175. PMID 12880493
- [Background] Simoni JM, Chen WT, Huh D, Fredriksen-Goldsen KI, Pearson C, Zhao H, Shiu CS, Wang X, Zhang F. A preliminary randomized controlled trial of a nurse-delivered medication adherence intervention among HIV-positive outpatients initiating antiretroviral therapy in Beijing, China. AIDS Behav. 2011 Jul;15(5):919-29. doi: 10.1007/s10461-010-9828-3. PMID 20957423
- [Background] Shet A, Arumugam K, Rodrigues R, Rajagopalan N, Shubha K, Raj T, D'souza G, De Costa A. Designing a mobile phone-based intervention to promote adherence to antiretroviral therapy in South India. AIDS Behav. 2010 Jun;14(3):716-20. doi: 10.1007/s10461-009-9658-3. PMID 20054634
- [Background] Konkle-Parker DJ, Erlen JA, Dubbert PM. Lessons learned from an HIV adherence pilot study in the Deep South. Patient Educ Couns. 2010 Jan;78(1):91-6. doi: 10.1016/j.pec.2009.04.010. Epub 2009 Jun 26. PMID 19560307
- [Background] Simoni JM, Pearson CR, Pantalone DW, Marks G, Crepaz N. Efficacy of interventions in improving highly active antiretroviral therapy adherence and HIV-1 RNA viral load. A meta-analytic review of randomized controlled trials. J Acquir Immune Defic Syndr. 2006 Dec 1;43 Suppl 1(0 1):S23-35. doi: 10.1097/01.qai.0000248342.05438.52. PMID 17133201
- [Background] Curioso WH, Kurth AE. Access, use and perceptions regarding Internet, cell phones and PDAs as a means for health promotion for people living with HIV in Peru. BMC Med Inform Decis Mak. 2007 Sep 12;7:24. doi: 10.1186/1472-6947-7-24. PMID 17850656
- [Background] Grant E, Logie D, Masura M, Gorman D, Murray SA. Factors facilitating and challenging access and adherence to antiretroviral therapy in a township in the Zambian Copperbelt: a qualitative study. AIDS Care. 2008 Nov;20(10):1155-60. doi: 10.1080/09540120701854634. PMID 19012078
- [Background] Murphy DA, Lu MC, Martin D, Hoffman D, Marelich WD. Results of a pilot intervention trial to improve antiretroviral adherence among HIV-positive patients. J Assoc Nurses AIDS Care. 2002 Nov-Dec;13(6):57-69. doi: 10.1177/1055329002238026. PMID 12469544
- [Background] Fisher JD, Fisher WA, Amico KR, Harman JJ. An information-motivation-behavioral skills model of adherence to antiretroviral therapy. Health Psychol. 2006 Jul;25(4):462-73. doi: 10.1037/0278-6133.25.4.462. PMID 16846321
- [Background] Holzemer WL, Henry SB, Portillo CJ, Miramontes H. The Client Adherence Profiling-Intervention Tailoring (CAP-IT) intervention for enhancing adherence to HIV/AIDS medications: a pilot study. J Assoc Nurses AIDS Care. 2000 Jan-Feb;11(1):36-44. doi: 10.1016/s1055-3290(06)60420-2. PMID 10670005
- [Background] Raney AA, Smith JK, Baker K. Adolescents and the appeal of video games. In P. Vorderer & J. Bryant (Eds.), Playing video games: Motives, responses and consequences. Mahwah, NJ: Lawrence Erlbaum 2006;165-180.
- [Background] Lee KM, Peng W. What do we know about social and psychological effects of computer games? A comprehensive review of the current literature. In P. Vorderer & J. Bryant (Eds.), Playing video games: Motives, responses and consequences (pp. 325-346). Mahwah, NJ: Lawrence Erlbaum 2006; 325-346.
- [Background] Starace F, Massa A, Amico KR, Fisher JD. Adherence to antiretroviral therapy: an empirical test of the information-motivation-behavioral skills model. Health Psychol. 2006 Mar;25(2):153-62. doi: 10.1037/0278-6133.25.2.153. PMID 16569106
- [Background] Fisher WA, Williams SS, Fisher JD, Malloy TE. Understanding AIDS risk behavior among sexually active urban adolescents: An empirical test of the information-motivation-behavioral skills model. AIDS and Behavior. 1999; 3:13-23.
- [Background] Fisher JD, Fisher WA, Misovich SJ, Kimble DL, Malloy TE. Changing AIDS risk behavior: effects of an intervention emphasizing AIDS risk reduction information, motivation, and behavioral skills in a college student population. Health Psychol. 1996 Mar;15(2):114-23. doi: 10.1037//0278-6133.15.2.114. PMID 8681919
- [Background] Bandura A.. Social foundations of thought and action: A Social cognitive theory. Englewood Cliffs, NJ: Prentice Hall, 1986.
- [Background] Lenhart A, Jones S, Macgill A. Adults and Video Games: A Pew Internet and American Life Study, December 2008 [Accessed on 8/13/13 : http://www.pewinternet.org/~/media//Files/Reports/2008/PIP_Adult_gaming_memo.pdf.pdf]
- [Background] Lieberman DA. Interactive video games for health promotion: Effects on knowledge, self-efficacy, social support, and health. In R.L. Street, W.R. Gold, & T. Manning (Eds.), Health promotion and interactive technology: Theoretical applications and future directions (pp. 103 120). Mahwah, NJ: Lawrence Erlbaum, 1997.
- [Background] Lieberman DA. What can we learn from playing interactive games? In P. Vorderer & J. Bryant (Eds.), Playing video games: Motives, responses and consequences (pp. 379-398).Mahwah, NJ: Lawrence Erlbaum, 2006.
- [Background] Paperny DM, Starn JR. Adolescent pregnancy prevention by health education computer games: computer-assisted instruction of knowledge and attitudes. Pediatrics. 1989 May;83(5):742-52. PMID 2654867
- [Background] Thomas R, Cahill J, Santilli L. Using an interactive computer game to increase skill and self-efficacy regarding safer sex negotiation: field test results. Health Educ Behav. 1997 Feb;24(1):71-86. doi: 10.1177/109019819702400108. PMID 9112099
- [Background] Homer C, Susskind O, Alpert HR, Owusu Ms, Schneider L, Rappaport LA, Rubin DH. An evaluation of an innovative multimedia educational software program for asthma management: report of a randomized, controlled trial. Pediatrics. 2000 Jul;106(1 Pt 2):210-5. PMID 10888694
- [Background] Brown SJ, Lieberman DA, Germeny BA, Fan YC, Wilson DM, Pasta DJ. Educational video game for juvenile diabetes: results of a controlled trial. Med Inform (Lond). 1997 Jan-Mar;22(1):77-89. doi: 10.3109/14639239709089835. PMID 9183781
- [Background] Shames RS, Sharek P, Mayer M, Robinson TN, Hoyte EG, Gonzalez-Hensley F, Bergman DA, Umetsu DT. Effectiveness of a multicomponent self-management program in at-risk, school-aged children with asthma. Ann Allergy Asthma Immunol. 2004 Jun;92(6):611-8. doi: 10.1016/S1081-1206(10)61426-3. PMID 15237762
- [Background] Cole SW, Kato PM, Marin-Bowling VM, Dahl GV, Pollock BH. Clinical trial of Re-Mission: A video game for young people with cancer. Cyberpsychology & Behavior. 2006; 9: 665-666.
- [Background] Kato PM, Cole SW, Bradlyn AS, Pollock BH. A video game improves behavioral outcomes in adolescents and young adults with cancer: a randomized trial. Pediatrics. 2008 Aug;122(2):e305-17. doi: 10.1542/peds.2007-3134. PMID 18676516
- [Background] Baranowski T, Buday R, Thompson DI, Baranowski J. Playing for real: video games and stories for health-related behavior change. Am J Prev Med. 2008 Jan;34(1):74-82. doi: 10.1016/j.amepre.2007.09.027. PMID 18083454
- [Background] Schunk DH. Vicarious influences on self-efficacy for cognitive skill learning. Journal of Social and Clinical Psychology. 1986;4 (3):316-327.
- [Background] Thompson D, Baranowski T, Buday R, Baranowski J, Thompson V, Jago R, Griffith MJ. Serious Video Games for Health How Behavioral Science Guided the Development of a Serious Video Game. Simul Gaming. 2010 Aug 1;41(4):587-606. doi: 10.1177/1046878108328087. PMID 20711522
- [Background] Wideman R, Owston R, Brown C, Kushniruk A, Ho F, Pitts K. Unpacking the potential of educational gaming: A new tool for gaming research. Simulation & Games: An International Journal. 2007;38:10-30.
- [Background] Stokes B. Video games have changed: Time to consider "serious games." The Development Education Journal. 2005. Retrieved August 20, 2011 from www.dea.org.uk.
- [Background] Brown LK, Lourie KJ, Pao M. Children and adolescents living with HIV and AIDS: a review. J Child Psychol Psychiatry. 2000 Jan;41(1):81-96. PMID 10763677
- [Background] Brown LK, Whiteley L, Peters A. HIV and AIDS. In The American Psychiatric Publishing Textbook of Child and Adolescent Psychiatry, Fourth Edition. (M. Dulcan, ed.), American Psychiatric Publishing, Inc. 2010; 32: 495-507.
- [Background] Whiteley LB, Brown LK, Swenson R, Kapogiannis BG, Harper GW. Disparities in mental health care among HIV-infected youth. J Int Assoc Provid AIDS Care. 2014 Jan-Feb;13(1):29-34. doi: 10.1177/2325957413488172. Epub 2013 May 21. PMID 23695228
- [Background] Brown LK, Schultz JR, Gragg RA. HIV-infected adolescents with hemophilia: adaptation and coping. The Hemophilia Behavioral Intervention Evaluation Project. Pediatrics. 1995 Sep;96(3 Pt 1):459-63. PMID 7651778
- [Background] Brown LK, Schultz JR, Parsons JT, Butler RB, Forsberg AD, Kocik SM, King G, Manco-Johnson M, Aledort L. Sexual behavior change among human immunodeficiency virus-infected adolescents with hemophilia. Adolescent Hemophilia Behavioral Intervention Evaluation Project Study Group. Pediatrics. 2000 Aug;106(2):E22. doi: 10.1542/peds.106.2.e22. PMID 10920178
- [Background] Nugent NR, Lally MA, Brown L, Knopik VS, McGeary JE. OPRM1 and diagnosis-related posttraumatic stress disorder in binge-drinking patients living with HIV. AIDS Behav. 2012 Nov;16(8):2171-80. doi: 10.1007/s10461-011-0095-8. PMID 22143634
- [Background] Whiteley LB, Brown LK, Swenson RR, Romer D, DiClemente RJ, Salazar LE, Vanable PA, Carey MP, Valois RF. African American adolescents and new media: associations with HIV/STI risk behavior and psychosocial variables. Ethn Dis. 2011 Spring;21(2):216-22. PMID 21749027
- [Background] Whiteley LB, Brown LK, Swenson RR, Valois RF, Vanable PA, Carey MP, DiClemente R, Salazar LF, Romer D. African American adolescents meeting sex partners online: closing the digital research divide in STI/HIV prevention. J Prim Prev. 2012 Feb;33(1):13-8. doi: 10.1007/s10935-012-0262-3. PMID 22293979
- [Background] Whiteley LB, Mello J, Hunt O, Brown LK. A review of sexual health web sites for adolescents. Clin Pediatr (Phila). 2012 Mar;51(3):209-13. doi: 10.1177/0009922811423311. Epub 2011 Sep 23. PMID 21946254
- [Background] Schuman P, Ohmit SE, Klein RS, Duerr A, Cu-Uvin S, Jamieson DJ, Anderson J, Shah KV; HIV Epidemiology Research Study (HERS) Group. Longitudinal study of cervical squamous intraepithelial lesions in human immunodeficiency virus (HIV)-seropositive and at-risk HIV-seronegative women. J Infect Dis. 2003 Jul 1;188(1):128-36. doi: 10.1086/375783. Epub 2003 Jun 17. PMID 12825181
- [Background] Cu-Uvin S, Hogan JW, Caliendo AM, Harwell J, Mayer KH, Carpenter CC; HIV Epidemiology Research Study. Association between bacterial vaginosis and expression of human immunodeficiency virus type 1 RNA in the female genital tract. Clin Infect Dis. 2001 Sep 15;33(6):894-6. doi: 10.1086/322613. Epub 2001 Aug 10. PMID 11512096
- [Background] Romero LM, Galbraith JS, Wilson-Williams L, Gloppen KM. HIV prevention among African American youth: how well have evidence-based interventions addressed key theoretical constructs? AIDS Behav. 2011 Jul;15(5):976-91. doi: 10.1007/s10461-010-9745-5. PMID 20635131
- [Background] Resnicow K, Dilorio CK, Davis R. Culture and development of HIV prevention and treatment programs. In Edgart, Noar SM, Freimuth, editors. Communication perspectives for Aids in the 21st Century pg 193-220.
- [Background] Bull SS, Phibbs S, Watson S, McFarlane M. What do young adults expect when they go online? Lessons for development of an STD/HIV and pregnancy prevention website. J Med Syst. 2007 Apr;31(2):149-58. doi: 10.1007/s10916-006-9050-z. PMID 17489508
- [Background] Romer D, Sznitman S, DiClemente R, Salazar LF, Vanable PA, Carey MP, Hennessy M, Brown LK, Valois RF, Stanton BF, Fortune T, Juzang I. Mass media as an HIV-prevention strategy: using culturally sensitive messages to reduce HIV-associated sexual behavior of at-risk African American youth. Am J Public Health. 2009 Dec;99(12):2150-9. doi: 10.2105/AJPH.2008.155036. Epub 2009 Oct 15. PMID 19833995
- [Background] Brown LK, DiClemente RJ, Beausoleil NI. Comparison of human immunodeficiency virus related knowledge, attitudes, intentions, and behaviors among sexually active and abstinent young adolescents. J Adolesc Health. 1992 Mar;13(2):140-5. doi: 10.1016/1054-139x(92)90081-l. PMID 1627582
- [Background] Lane SJ, Heddle NM, Arnold E, Walker I. A review of randomized controlled trials comparing the effectiveness of hand held computers with paper methods for data collection. BMC Med Inform Decis Mak. 2006 May 31;6:23. doi: 10.1186/1472-6947-6-23. PMID 16737535
- [Background] Lester RT, Ritvo P, Mills EJ, Kariri A, Karanja S, Chung MH, Jack W, Habyarimana J, Sadatsafavi M, Najafzadeh M, Marra CA, Estambale B, Ngugi E, Ball TB, Thabane L, Gelmon LJ, Kimani J, Ackers M, Plummer FA. Effects of a mobile phone short message service on antiretroviral treatment adherence in Kenya (WelTel Kenya1): a randomised trial. Lancet. 2010 Nov 27;376(9755):1838-45. doi: 10.1016/S0140-6736(10)61997-6. Epub 2010 Nov 9. PMID 21071074
- [Background] Johnson AM, Copas AJ, Erens B, Mandalia S, Fenton K, Korovessis C, Wellings K, Field J. Effect of computer-assisted self-interviews on reporting of sexual HIV risk behaviours in a general population sample: a methodological experiment. AIDS. 2001 Jan 5;15(1):111-5. doi: 10.1097/00002030-200101050-00016. PMID 11192852
- [Background] Balfour L, Kowal J, Tasca GA, Cooper CL, Angel JB, Macpherson PA, Garber G, Beique L, Cameron DW. Development and psychometric validation of the HIV Treatment Knowledge Scale. AIDS Care. 2007 Oct;19(9):1141-8. doi: 10.1080/09540120701352241. PMID 18058398
- [Background] Simoni JM, Kurth AE, Pearson CR, Pantalone DW, Merrill JO, Frick PA. Self-report measures of antiretroviral therapy adherence: A review with recommendations for HIV research and clinical management. AIDS Behav. 2006 May;10(3):227-45. doi: 10.1007/s10461-006-9078-6. PMID 16783535
- [Background] Stott NC, Rollnick S, Rees MR, Pill RM. Innovation in clinical method: diabetes care and negotiating skills. Fam Pract. 1995 Dec;12(4):413-8. doi: 10.1093/fampra/12.4.413. PMID 8826057
- [Background] Parsons JT, Rosof E, Mustanski B. Patient-related factors predicting HIV medication adherence among men and women with alcohol problems. J Health Psychol. 2007 Mar;12(2):357-70. doi: 10.1177/1359105307074298. PMID 17284499
- [Background] Davies G, Koenig LJ, Stratford D, Palmore M, Bush T, Golde M, Malatino E, Todd-Turner M, Ellerbrock TV. Overview and implementation of an intervention to prevent adherence failure among HIV-infected adults initiating antiretroviral therapy: lessons learned from Project HEART. AIDS Care. 2006 Nov;18(8):895-903. doi: 10.1080/09540120500329556. PMID 17012078
- [Background] Derogatis L, Spencer M. The Brief Symptom Inventory (BSI): Administration, scoring, and procedures manual-1. Baltimore: Johns Hopkins University School of Medicine, Clinical Psychometrics Research Unit, 1982.
- [Background] WHO ASSIST Working Group. The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST): development, reliability and feasibility. Addiction. 2002 Sep;97(9):1183-94. doi: 10.1046/j.1360-0443.2002.00185.x. PMID 12199834
- [Background] Brown LK, Hadley W, Stewart A, Lescano C, Whiteley L, Donenberg G, DiClemente R; Project STYLE Study Group. Psychiatric disorders and sexual risk among adolescents in mental health treatment. J Consult Clin Psychol. 2010 Aug;78(4):590-7. doi: 10.1037/a0019632. PMID 20658815
- [Background] Raudenbush S, Bryk A. Hierarchical Linear Models (Second Edition). Thousand Oaks: Sage Publications, 2002.
- [Background] Raudenbush S, Bryk A. Applied Longitudinal Data Analysis. Singer & Willett, 2003.
- [Background] Kraemer HC, Mintz J, Noda A, Tinklenberg J, Yesavage JA. Caution regarding the use of pilot studies to guide power calculations for study proposals. Arch Gen Psychiatry. 2006 May;63(5):484-9. doi: 10.1001/archpsyc.63.5.484. PMID 16651505
- [Background] Spybrook J, Raudenbush SW, Liu X-feng, Congdon R, Martinez A. Optimal design for Longitudinal and Multilevel Research: Documentation for the "Optimal Design" Software, 2008.
- [Background] Brown LK, Nugent NR, Houck CD, Lescano CM, Whiteley LB, Barker D, Viau L, Zlotnick C. Safe Thinking and Affect Regulation (STAR): human immunodeficiency virus prevention in alternative/therapeutic schools. J Am Acad Child Adolesc Psychiatry. 2011 Oct;50(10):1065-74. doi: 10.1016/j.jaac.2011.06.018. Epub 2011 Aug 27. PMID 21961780
- [Background] Dixon EE, Whiteley L, Curtis V, Beausoleil N, Brown LK. Attitudes About Pre-Exposure Prophylaxis Among Urban Minority Youth: Associations With Sexual and Substance Use Behaviors. Presented at the Annual meeting of the American Academy of Child and Adolescent Psychiatry, Orlando, FL; October 22-27, 2013.
- [Background] Whiteley L, Brown LK, Curtis V, Heck N. An iPhone App/Game to Improve ART Adherence. To be presented at the 9th International Conference on HIV Treatment and Prevention Adherence, Miami, FL; June 8-10, 2014.
- [Background] Hosek SG, Siberry G, Bell M, Lally M, Kapogiannis B, Green K, Fernandez MI, Rutledge B, Martinez J, Garofalo R, Wilson CM; Adolescent Trials Network for HIVAIDS Interventions (ATN). The acceptability and feasibility of an HIV preexposure prophylaxis (PrEP) trial with young men who have sex with men. J Acquir Immune Defic Syndr. 2013 Apr 1;62(4):447-56. doi: 10.1097/QAI.0b013e3182801081. PMID 24135734
- [Background] Fisher JD, Fisher WA, Shuper PA. The Information-Motivation-Behavioral Skills Model of HIV preventive behavior. In R. DiClemente, R. Crosby, & M. Kegler (Eds.), Emerging theories in health promotion practice and research model of HIV preventive behavior. (2nd ed., pp. 22-63). San Francisco, CA: Jossey Bass Publishers 2009.
- [Background] Fisher JD, Amico KR, Fisher WA, Harman JJ. The information-motivation-behavioral skills model of antiretroviral adherence and its applications. Curr HIV/AIDS Rep. 2008 Nov;5(4):193-203. doi: 10.1007/s11904-008-0028-y. PMID 18838059
- [Background] Fisher WA, Fisher JD, Harman J. The information-motivation-behavioral skills model: A general social psychological approach to understanding and promoting health behavior. In J. Suls, & K. A. Wallston (Eds.), Social psychological foundations of health and illness (pp. 82-106). United Kingdom: Blackwell Publishers, 2003.
- [Background] Fisher JD, Fisher WA, Bryan AD, Misovich SJ. Information-motivation-behavioral skills model-based HIV risk behavior change intervention for inner-city high school youth. Health Psychol. 2002 Mar;21(2):177-86. PMID 11950108
- [Background] Bachman Desilva M, Gifford AL, Keyi X, Li Z, Feng C, Brooks M, Harrold M, Yueying H, Gill CJ, Wubin X, Vian T, Haberer J, Bangsberg D, Sabin L. Feasibility and Acceptability of a Real-Time Adherence Device among HIV-Positive IDU Patients in China. AIDS Res Treat. 2013;2013:957862. doi: 10.1155/2013/957862. Epub 2013 Jul 16. PMID 23956851
- [Background] Haberer JE, Kahane J, Kigozi I, Emenyonu N, Hunt P, Martin J, Bangsberg DR. Real-time adherence monitoring for HIV antiretroviral therapy. AIDS Behav. 2010 Dec;14(6):1340-6. doi: 10.1007/s10461-010-9799-4. PMID 20809380
- [Background] Anderson PL, Kiser JJ, Gardner EM, Rower JE, Meditz A, Grant RM. Pharmacological considerations for tenofovir and emtricitabine to prevent HIV infection. J Antimicrob Chemother. 2011 Feb;66(2):240-50. doi: 10.1093/jac/dkq447. Epub 2010 Nov 30. PMID 21118913

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Subjects in the intervention group will each receive smartphones with a data service plan. The IMB Gaming Intervention is designed to improve information, motivation, and skills about adherence and HIV preventative behaviors throughout play. The mission of Viral Combat is: kill virus and build strength through taking medicine, learning HIV prevention information, and engaging with healthy characters in order to improve motivation and build skills. Participants will get a game graphic with a supportive message such as "Missing you: Get in the Game" to their phones. Throughout the gaming intervention subjects will continue routine clinical care visits and HIV testing in the PrEP clinic.
  IMB Gaming Intervention
Period: Overall Study
Arm/Group | Intervention | Comparison
Started | 41 | 41
Immediate Posttest (3 Months) | 33 | 34
6-month Follow-up | 32 | 35
Completed | 32 | 35
Not Completed | 9 | 6
Not completed — Withdrawal by Subject | 7 | 2
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Intervention: The IMB Gaming Intervention is designed to improve information, motivation, and skills about adherence and HIV preventative behaviors throughout play. The mission of Viral Combat is: kill virus and build strength through taking medicine, learning HIV prevention information, and engaging with healthy characters in order to improve motivation and build skills. Participants will get a game graphic with a supportive message such as "Missing you: Get in the Game" to their phones. Throughout the gaming intervention subjects will continue routine clinical care visits and HIV testing in the PrEP clinic.
  IMB Gaming Intervention
- Total: Total of all reporting groups
Arm/Group | Intervention | Comparison | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.8 (4.4) | 24.8 (3.9) | 24.8 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 40 | 41 | 81
    Female | 0 | 3 | 3
    Male | 40 | 38 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 39 | 39 | 78
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 36 | 70
  White | 4 | 3 | 7
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1
Insurance Type [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 40 | 41 | 81
    None | 8 | 8 | 16
    Public | 10 | 11 | 21
    Private | 22 | 22 | 44
Time on PrEP [Count of Participants; unit: Participants]
  Less than one month | 9 | 6 | 15
  One month or more | 32 | 35 | 67
Sexual Orientation [Count of Participants; unit: Participants]
  Heterosexual | 1 | 0 | 1
  Homosexual | 27 | 29 | 56
  Bisexual | 13 | 12 | 25
Health Literacy [Count of Participants; unit: Participants] — Item: "How often do you need to have someone help you when you read instructions, pamphlets, or other written materials from your doctor or pharmacy?". Participants respond on a 5-point scale of "Never" to "Always".
  Participants
    Never | 26 | 32 | 58
    Rarely | 11 | 6 | 17
    Sometimes | 4 | 3 | 7
    Often | 0 | 0 | 0
    Always | 0 | 0 | 0
Global Severity Index [Mean (Standard Deviation); unit: units on a scale] — Psychological distress was assessed by the Global Symptom Index of the 18-item Brief Symptom Inventory (BSI-18). Response options ranged from 0 (Never) to 4 (Extremely). Higher scores indicate greater experienced psychological distress.
  units on a scale | 0.5 (0.8) | 0.3 (0.8) | 0.4 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Self-Report of PrEP Adherence
Description: Self-report measure of adherence in the past 7 days categorized as "optimal" (0-3 missed doses in the past 7 days) versus "suboptimal" (4-7 missed doses in the past 7 days).
Time Frame: 24 weeks
Population: Loss to follow-up, withdrawals, and missing data account for the discrepancy in the analysis population.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Subjects in the intervention group will each receive a smartphone with a data service plan. The IMB Gaming Intervention is designed to improve information, motivation, and skills about adherence and HIV preventative behaviors throughout play. The mission of Viral Combat is: kill virus and build strength through taking medicine, learning HIV prevention information, and engaging with healthy characters in order to improve motivation and build skills. Participants will get a game graphic with a supportive message such as "Missing you: Get in the Game" to their phones. Throughout the gaming intervention subjects will continue routine clinical care visits and HIV testing in the PrEP clinic.
  IMB Gaming Intervention
Arm/Group | Intervention | Comparison
Number analyzed (Participants) | 31 | 34
Participants
  Optimal adherence | 22 | 26
  Suboptimal adherence | 9 | 8

2. Primary Outcome: ARV (TFV-DP) Levels
Description: Intracellular TFV-DP will be measured in red blood cells using dried blood spots. TFV-DP levels provide a measure of long-term adherence over the preceding month (like hemoglobin A1C). The level of intracellular TFV-DP can be used to estimate how many doses/week the participant is taking on average (e.g. 7/wk on average, 4-7/wk on average, 2-4/wk on average, <2/wk on average).
Time Frame: 24 weeks
Population: Missing data, withdrawals, and those lost to follow-up account for the discrepancy in the analysis population.
Measure: Mean (Standard Deviation); unit: fmol/punch
Groups:
- Intervention: Subjects in the intervention will each receive a smartphone with a data service plan. The IMB Gaming Intervention is designed to improve information, motivation, and skills about adherence and HIV preventative behaviors throughout play. The mission of Viral Combat is: kill virus and build strength through taking medicine, learning HIV prevention information, and engaging with healthy characters in order to improve motivation and build skills. Participants will get a game graphic with a supportive message such as "Missing you: Get in the Game" to their phones. Throughout the gaming intervention subjects will continue routine clinical care visits and HIV testing in the PrEP clinic.
  IMB Gaming Intervention
Arm/Group | Intervention | Comparison
Number analyzed (Participants) | 27 | 28
fmol/punch | 810.4 (662.6) | 574.6 (668.9)

3. Secondary Outcome: HIV Knowledge at 24 Weeks
Description: The HIV Knowledge Scale assesses knowledge about issues such as risks for HIV, using 5 items with "true," "false," or "do not know" response options. Total scores range from 0 to 5. Higher scores indicate greater knowledge.
Time Frame: 24 weeks
Population: Missing data, withdrawals, and loss to follow-up account for the discrepancy in the analysis population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Comparison
Number analyzed (Participants) | 31 | 34
units on a scale | 4.1 (1.1) | 4.2 (1.1)

4. Secondary Outcome: Motivational Readiness for Adherence at 24 Weeks
Description: Rollnick's Readiness Ruler will be used to assess motivation for adherence to medication and medical visits. Respondents rate how ready they are to take PrEP as prescribed on a scale from 1 (not ready) to 10 (ready to be consistent or already consistent) each month.
Time Frame: 24 weeks
Population: Missing data, withdrawals and loss to follow-up account for the discrepancy in the analysis population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Comparison
Number analyzed (Participants) | 31 | 34
units on a scale | 9.1 (2.4) | 9.8 (0.6)

5. Other Pre Specified Outcome: Social Support for Medication Adherence
Description: This six item measure assesses social support for taking medications, going to medical appointments and other tasks related to adherence using Likert style items with a four point scale. Scores range from 6 to 24 Higher scores indicate greater social support.
Time Frame: 24 weeks
Population: Missing data, withdrawals and loss to follow-up accounts for the discrepancy in the analysis population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Comparison
Number analyzed (Participants) | 31 | 34
units on a scale | 21.4 (3.9) | 21.2 (5.4)

6. Primary Outcome: Average Number of Days on PrEP Per Week
Description: The level of intracellular TFV-DP can be used to estimate how many doses/week the participant is taking on average in the past month (e.g. 7/wk on average, 4-7/wk on average, 2-4/wk on average, <2/wk on average).
Time Frame: 24 weeks
Population: Missing data, withdrawals, and those lost to follow-up account for the discrepancy in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Comparison
Number analyzed (Participants) | 27 | 28
Participants
  Undetectable levels | 5 | 6
  Less than 2 days (<350 fmol/punch) | 4 | 7
  2-3 days (350-699 fmol/punch) | 3 | 8
  4-6 days (700-1249 fmol/punch) | 7 | 2
  7 days (greater than or equal to 1250 fmol/punch) | 8 | 5

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 24 weeks.
Description: Adverse events as described in the study protocol were reported by study staff to the principle investigator.
Arm/Group | Intervention | Comparison
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 0/41

LIMITATIONS AND CAVEATS:
This study had a small sample. Participants were recruited from Jackson, MS, so this sample is not nationally representative. Self-reported adherence data is subject to social desirability bias. Intervention app was only available for iPhone users.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT02611362/Prot_SAP_000.pdf